CLINICAL TRIAL: NCT06665815
Title: A National Screening Program for Islet Autoantibodies Among First-degree Relatives of T1D Patients
Acronym: ADIR Families
Status: Recruiting | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0483-24RMC
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes; Autoantibodies Screening
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Negative result at the autoantibodies screening test: 1. Participants without positive autoantibodies will not be confirmed or referred to follow up
  2. Participants with only one positive autoantibody, will be referred to perform regular follow up as part of routine medical care according to the international consensus guidelines published in July 2024
- Positive result at the autoantibodies screening test: Participants with two or more positive autoantibodies:
  1. will be invited to perform a confirmation test as part of the study
  2. If confirmed as having pre-symptomatic type 1 diabetes (T1D) (stages 1 / 2), participants will be referred to complete an educational program emphasizing on DKA prevention and to perform regular follow-up according to the international consensus guidelines published in July 2024, as part of routine medical care

SUMMARY:
A national Screening program for the presence of Islet Autoantibodies (IA) in relatives of people with type 1 diabetes (PWT1D) aiming at identifying people with pre-clinical (stage 1 & 2) T1D and DKA prevention on the clinical presentation of T1D. All participants will be screened at study entry for the presence of 4 islet autoantibodies: glutamic acid decarboxylase antibody (GADA), insulinoma-associated-2 antibody (IA-2A), insulin antibodies (IAA) and Zinc transporter-8 antibodies (ZnT8A). The ADAP assay will be used to detect IA.

A confirmation blood sample for positive participants with two or more IA will be taken. The confirmation analysis will be done by the ADAP assay, conventional ELISA, and RIA.

Participants identified as part of the study with pre-symptomatic type 1 diabetes (T1D) (stages 1 and 2) will be referred to complete an educational program emphasizing DKA prevention as part of routine medical care .During the study, cases of stage 2 and stage 3 diabetes and DKA events in participants who are positive for IA will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-45 years
* First-degree relatives of Type 1 Diabetes probands
* Signing an informed consent

Exclusion Criteria:

* Known diabetes of any kind (type 1, type 2, MODY)
* Have a previous history of being treated with insulin or oral diabetes medications.
* Currently, using systemic immunosuppressive agents (topical and inhaled agents are acceptable)

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: First degree relatives of patients with Type 1 diabetes from all over Israel, aged 2-45 years old
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
The prevalence of multiple antibodies among first-degree relatives of Type I Diabetes probands in Israel | End of screening, 3 years after obtaining the first screening test

SECONDARY OUTCOMES:
The prevalence of Diabetic Ketoacidosis at Type 1 Diabetes presentation among the screened cohort | End of screening, 3 years after obtaining the first screening test
Proportion and rate of progression from stage 1 to stage 2 and stage 3 Type 1 Diabetes | End of screening, 3 years after obtaining the first screening test
>500 individuals with pre-clinical Type 1 Diabetes identified in the cohort | End of screening, 3 years after obtaining the first screening test

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof., Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Children Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No